CLINICAL TRIAL: NCT04596319
Title: A Phase 1b/2a, Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety and Tolerability of AP-PA02 Multi-Phage Therapeutic Candidate for Inhalation in Subjects With Cystic Fibrosis and Chronic Pulmonary Pseudomonas Aeruginosa (Pa) Infection
Brief Title: Ph 1/2 Study Evaluating Safety and Tolerability of Inhaled AP-PA02 in Subjects With Chronic Pseudomonas Aeruginosa Lung Infections and Cystic Fibrosis
Acronym: SWARM-Pa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP-PA02-101
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa; Pseudomonas; Lung Infection; Lung Infection Pseudomonal
Keywords: phage; bacteriophage; cystic fibrosis; Pseudomonas; Pseudomonas aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AP-PA02 (Experimental): Anti-pseudomonal bacteriophage
  Interventions: Biological: AP-PA02
- Placebo (Placebo Comparator): Inactive isotonic solution
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AP-PA02 — Bacteriophage administered via inhalation
  Arms: AP-PA02
Other: Placebo — Inactive Placebo administered via inhalation
  Arms: Placebo

SUMMARY:
Phase 1b/2a, double-blind, randomized, placebo-controlled, single and multiple ascending dose study to evaluate the safety, tolerability and phage recovery profile of AP-PA02 multi-bacteriophage therapeutic candidate administered by inhalation in subjects with cystic fibrosis and chronic pulmonary Pseudomonas aeruginosa (PA) infection.

DETAILED DESCRIPTION:
The study consists of two parts. Subjects with Cystic Fibrosis and chronic pulmonary Pseudomonas aeruginosa (PA) infection will be enrolled in either Part 1 (single-ascending dose cohorts) or Part 2 (multiple-ascending dose cohorts).

Part 1 will evaluate single doses of AP-PA02 at two ascending dose levels, administered by inhalation. Treatment assignment will be randomized, double-blind, placebo-controlled in each of two ascending dose cohorts. Part 2 will also be double-blinded, randomized, placebo controlled, and will evaluate the safety and efficacy of multiple doses of AP-PA02 in each of two ascending dose level cohorts.

Subjects in both Parts 1 and 2 will be followed for approximately 4 weeks and evaluated for safety, tolerability, phage titer profile and immunogenicity.

ELIGIBILITY:
Key Inclusion Criteria:

* ≥ 18 years old
* Body mass index (BMI) of ≥ 18 kg/m2
* Documented diagnosis of CF
* Evidence of chronic pulmonary Pseudomonas aeruginosa infection
* Willing to undergo sputum induction procedures at designated study visits, and willing to provide expectorated sputum samples at all other timepoints (for subjects who are able to expectorate)
* For SAD: FEV1 ≥ 60% of predicted normal [per Global Lung Function Initiative (GLI) standards] at Screening
* For MAD: FEV1 ≥ 40% of predicted normal [per Global Lung Function Initiative (GLI) standards] at Screening
* Adequate renal function

Key Exclusion Criteria:

* Recent significant weight loss
* Abnormal vital signs at Screening
* History of prolonged QT syndrome
* Use of supplemental oxygen during the day at rest
* Abnormal liver function tests greater than 3X the upper limit of normal (ULN)
* Recent oral or IV antibiotics received for acute pulmonary exacerbation. Inhaled antibiotic use for chronic suppression of P. aeruginosa is acceptable.
* Recent clinically significant infection requiring systemic antimicrobial therapy
* Currently receiving anti-pseudomonal antibiotic treatment for acute sinusitis.
* Currently receiving systemic corticosteroids
* Currently receiving treatment for active infection with nontuberculous mycobacteria (NTM), Staphylococcus aureus, or Burkholderia cepacia complex lung infection
* Currently receiving treatment for aspergillosis or ABPA (allergic bronchopulmonary aspergillosis)
* Initiation of a CFTR potentiator/corrector therapy, such as Trikafta®, less than 90 days prior to Screening
* Acquired or primary immunodeficiency syndromes
* Active pulmonary malignancy (primary or metastatic)
* History of lung transplantation
* Recent hemoptysis
* Female pregnant or breastfeeding
* Heavy smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mina Pastagia, MD, MS, Study Director — Armata Pharmaceuticals, Inc.
Locations (20):
- United States (20):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - St. Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Harper University Hospital, Detroit, Michigan
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New York Medical College, Valhalla, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Armata Pharmaceuticals, Inc. — http://armatapharma.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Percentages were based on the number of subjects in the Safety Population in each treatment group. The Safety Population included all subjects who were administered at least 1 dose of study treatment.
Groups:
- Cohort 1 SAD: 3-phage (1x10^10 PFU single dose)
- Cohort 2 SAD: 3-phage (3x10^10 PFU single dose)
- Amendment 5 MAD: 3-phage multiple ascending dose (1E10 PFU/dose x3 doses/day x 3 days)
- Cohort 3 MAD: 5-phage (5.75x10^10 PFU/dose x 2 doses/day x 5 days)
- Cohort 4 MAD: 5-phage (1.5x10^11 PFU/dose x 2 doses/day x 10 days)
- SAD Placebo: Single dose placebo
- MAD Placebo: Multiple ascending dose placebo
Period: Overall Study
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Amendment 5 MAD | Cohort 3 MAD | Cohort 4 MAD | SAD Placebo | MAD Placebo
Started | 3 | 3 | 2 | 3 | 10 | 3 | 5
Completed | 3 | 3 | 2 | 3 | 10 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Amendment 5 MAD: 3-phage (1E10 PFU/dose x 3 doses/day x 3 days)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Amendment 5 MAD | Cohort 3 MAD | Cohort 4 MAD | SAD Placebo | MAD Placebo | Total
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 10 | 3 | 5 | 29
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at screening | 41.7 (3.21) | 40.7 (6.03) | 31.5 (9.5) | 44.3 (18.72) | 38.2 (8.65) | 39.6 (19.36) | 47.8 (16.15) | 40.8 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 2 | 6 | 2 | 1 | 16
  Male | 1 | 0 | 2 | 1 | 4 | 1 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 2 | 3 | 10 | 3 | 5 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 2 | 3 | 10 | 3 | 4 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity Treatment Emergent Adverse Events (TEAEs)
Description: Incidence and severity of treatment emergent adverse events of single and multiple doses of AP-PA02 administered by inhalation
Time Frame: Day 1 pre-dose through End of Study Visit (28 days post last dose of study drug), up to 4 weeks for single ascending dose and up to 5.5 weeks for multiple ascending dose.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: 3-phage (1x10^10 PFU single dose)
- Cohort 2: 3-phage (3x10^10 PFU single dose)
- Amendment 5: 3-phage multiple ascending dose (1E10 PFU/dose x3 doses/day x 3 days)
- Cohort 3: 5-phage (5.75x10^10 PFU/dose x 2 doses/day x 5 days)
- Cohort 4: 5-phage (1.5x10^11 PFU/dose x 2 doses/day x 10 days)
- MAD Placebo: multiple dose placebo
Arm/Group | Cohort 1 | Cohort 2 | Amendment 5 | Cohort 3 | Cohort 4 | SAD Placebo | MAD Placebo
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 10 | 3 | 5
Participants
  Any TEAEs | 1 | 1 | 1 | 0 | 5 | 2 | 4
  Any serious TEAEs | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Any IMP-related TEAEs | 0 | 0 | 0 | 0 | 4 | 0 | 2
  Any IMP-related serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAEs with Grade 1 (mild) as the worst severity | 0 | 0 | 0 | 0 | 4 | 2 | 2
  Any TEAEs with Grade 2 (moderate) as the worst severity | 1 | 1 | 1 | 0 | 0 | 1 | 2
  Any TEAEs with Grade 3 (severe) as the worst severity | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Any TEAEs with Grade 4 (life-threatening) as the worst severity | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAEs with Grade 5 (death) as the worst severity | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 pre-dose through End of Study Visit (28 days post last dose of study drug), up to 4 weeks for single ascending dose and up to 5.5 weeks for multiple ascending dose
Description: Adverse events were coded using MedDRA Version 23.0. At each level of summarization, subjects who experienced more than 1 event were counted only once.
Arm/Group | Cohort 1 SAD | Cohort 2 SAD | Amendment 5 MAD | Cohort 3 MAD | Cohort 4 MAD | SAD Placebo | MAD Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/3 | 0/10 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/3 | 1/10 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/2 | 0/3 | 5/10 | 2/3 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 SAD (N=3) | Cohort 2 SAD (N=3) | Amendment 5 MAD (N=2) | Cohort 3 MAD (N=3) | Cohort 4 MAD (N=10) | SAD Placebo (N=3) | MAD Placebo (N=5)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 SAD (N=3) | Cohort 2 SAD (N=3) | Amendment 5 MAD (N=2) | Cohort 3 MAD (N=3) | Cohort 4 MAD (N=10) | SAD Placebo (N=3) | MAD Placebo (N=5)
chills (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1
sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2
trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Backache (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publications policy is also provided in the Clinical Trial Agreement. The data from this study will be available to the Investigators for publication upon the completion of the study. The Sponsor agrees to have the results published, whether positive or negative. The Sponsor will review any manuscripts to ensure that proprietary information has the appropriate patent protection prior to journal submission.

DOCUMENTS (2):
  • Study Protocol (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT04596319/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT04596319/SAP_001.pdf